CLINICAL TRIAL: NCT02065817
Title: Dose of Labeled Cholesterol and Phenylalanine for HDL Kinetics: A Pilot Study
Brief Title: Dose of Labeled Cholesterol for Kinetics: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ananda Basu, PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13-004890
Record Dates: First submitted 2014-02-13; First posted 2014-02-19 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Lipid Metabolism
Keywords: Lipid; Apolipoproteins; Cardiovascular disease risks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tracer (Experimental)
  Interventions: Other: stable isotope of cholesterol

INTERVENTIONS:
Other: stable isotope of cholesterol

SUMMARY:
This is a pilot study to determine the optimum time and dose to draw blood samples using a tracer for HDL kinetics.

ELIGIBILITY:
Inclusion Criteria:

• Healthy men and women ages 18 - 50

Exclusion Criteria:

* Cardiovascular disease
* Metabolic disease
* Hematologic disorder
* Liver or kidney disease
* phenylketonuria
* Currently taking lipid lowering medications or any other drugs that could affect lipid metabolism

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2014-02; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Incorporation of orally administered 13C3 cholesterol into plasma cholesterol | 72 hours
  13C3 cholesterol, which is labeled with a stable isotope, will be administered orally. Blood samples will be taken every 4-6 hours for 72 hours for the measurement of stable isotopic enrichment in cholesterol using gas chromatography-mass spectrometry. The study has a dual purpose: to determine the optimum oral dose of isotope, and to determine the time of peak enrichment in plasma cholesterol.

CONTACTS AND LOCATIONS:
Overall Officials: John M Miles, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States